CLINICAL TRIAL: NCT01309607
Title: Phase II Open-Label Study of Preoperative Weekly Paclitaxel and Carboplatin With Lapatinib (Tykerb®) in Patients With ErbB2-Positive Stage I-III Breast Cancer
Brief Title: Study of Preoperative Weekly Paclitaxel and Carboplatin With Lapatinib (Tykerb®) in Patients With ErbB2-Positive Stage I-III Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR07/29/10
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: ErbB2-Positive Stage I-III Breast Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre-operative Therapy (Experimental): Neoadjuvant paclitaxel/carboplatin/lapatinib x 12 weeks
  Interventions: Drug: paclitaxel/carboplatin/lapatinib

INTERVENTIONS:
Drug: paclitaxel/carboplatin/lapatinib — Drug doses for the neoadjuvant regimen:
  * Paclitaxel 80mg/m2, day 1, 8, 15 of a 21-day cycle
  * Carboplatin AUC of 2, day 1, 8 of a 21-day cycle
  * Lapatinib 750mg daily continuously

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of weekly paclitaxel and carboplatin, in combination with lapatinib, in the neoadjuvant treatment of non-metastatic erbB2-positive breast cancer.

Secondary objectives include:

* To determine the safety and tolerability of weekly paclitaxel and carboplatin, combined with lapatinib, in an Asian population
* To determine breast conservation rates following neoadjuvant paclitaxel/ carboplatin/ lapatinib
* To determine clinical response rates and relapse-free survival of patients treated with neoadjuvant paclitaxel/ carboplatin/ lapatinib
* To identify predictive tumour biomarkers for pathologic complete response

The investigators hypothesize that pathologic complete response rates will be improved from 15% to 35% with the neoadjuvant regimen of carboplatin/ paclitaxel/ lapatinib compared to standard chemotherapy alone in HER2 positive early stage breast cancers.

DETAILED DESCRIPTION:
* Pathologic complete response following neoadjuvant chemotherapy has been shown to be an independent, strong predictor of disease-free and overall survival in operable breast cancer
* The addition of neoadjuvant trastuzumab to chemotherapy results in a 2-3 fold increase in pCR rates in operable ErbB2-positive breast cancer
* Lapatinib is being explored as an alternative to trastuzumab in large clinical trials in operable ErbB2-positive breast cancer
* In a randomised phase III adjuvant trial, BCIRG 006, non-anthracycline chemotherapy (docetaxel and carboplatin) has been shown to be as effective as conventional sequential anthracycline-containing chemotherapy and docetaxel, in combination with trastuzumab, but with improved cardiac safety
* Weekly paclitaxel has been shown in a randomized phase III study to be the optimal adjuvant taxane regimen
* Weekly paclitaxel and carboplatin, in combination with lapatinib, has demonstrated safety and efficacy in Phase I/II clinical studies of metastatic breast and ovarian cancer
* The investigators aim to assess the efficacy of a non-anthracycline containing regimen, weekly paclitaxel and carboplatin, in combination with lapatinib in inducing pCR in the neoadjuvant treatment of ErbB2-positive non-metastatic breast cancer. The investigators hypothesize that this combination will achieve pCR rates of at least 35%

ELIGIBILITY:
Inclusion Criteria:

* • Female, Age ≥ 18 years

  * Histologic or cytologic diagnosis of breast carcinoma
  * T1-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with the largest diameter measuring 2.0cm or greater by calipers
  * Tumor is HER2 positive either by IHC (3+) or FISH amplification (amplification ratio >2.2)
  * Patients must not have received prior chemotherapy or hormonal therapy for the treatment of breast cancer
  * Karnofsky performance status of 70 or higher
  * Estimated life expectancy of at least 12 weeks
  * Adequate organ function including the following:

Bone marrow:

* Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L
* Platelets >= 100 x 109/L

Hepatic:

* Bilirubin <= 1.5 x upper limit of normal (ULN),
* ALT or AST <= 2.5x ULN

Renal:

o Calculated creatinine clearance >30ml/minute

* Left ventricular ejection fraction >=50% measured by 2D echo or MUGA
* Signed informed consent from patient or legal representative
* Patient with reproductive potential must use an approved contraceptive method if appropriate (e.g. intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment

Exclusion Criteria:

* • Prior treatment for locally advanced or metastatic breast cancer

  * Treatment within the last 30 days with any investigational drug
  * Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy
  * Major surgery within 28 days of study drug administration
  * Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
  * Breast feeding
  * Serious cardiac illness or medical conditions including but not confined to:

    * History of documented congestive cardiac failure or systolic dysfunction (LVEF <50%)
    * High-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV block, supraventricular arrhythmias which are not adequately rate-controlled)
    * History of significant ischaemic heart disease
    * Clinically significant valvular heart disease
    * Poorly controlled hypertension (e.g. systolic BP > 180mmHg or diastolic >100mmHg)
  * Poorly controlled diabetes mellitus.
  * Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
  * History of significant neurological or mental disorder, including seizures or dementia.
  * Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones or stable chronic liver disease per investigator assessment)
  * Concomitant use of CYP3A4 inhibitors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of pathologic complete response | 12 weeks

SECONDARY OUTCOMES:
Treatment related toxicities | 12 weeks
Breast conservation rates | 16 weeks
Clinical response rates | 1 year
Relapse free survival (RFS) | 2 years
Identification of tumor biomarkers that predict pathologic complete response | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 1998 Aug;16(8):2672-85. doi: 10.1200/JCO.1998.16.8.2672. PMID 9704717
- [Background] Geyer CE, Forster J, Lindquist D, Chan S, Romieu CG, Pienkowski T, Jagiello-Gruszfeld A, Crown J, Chan A, Kaufman B, Skarlos D, Campone M, Davidson N, Berger M, Oliva C, Rubin SD, Stein S, Cameron D. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006 Dec 28;355(26):2733-43. doi: 10.1056/NEJMoa064320. PMID 17192538